CLINICAL TRIAL: NCT04623112
Title: Do Severe-profound Hearing Impaired Adults Perform Better in Speech Perception With Frequency Compression Switched on or Off or Fitted to Hearing Loss
Brief Title: Use of Frequency Compression in Severe-profound Hearing Loss Adults
Acronym: FC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/0217
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Frequency Compression; Severe-profound Hearing Impairment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- FC Deactivated (Other): Frequency Compression feature on hearing aids is deactivated for 4 weeks
  Interventions: Device: Hearing aid feature: Frequency Compression
- FC activated & set to default (Experimental): Frequency compression feature activated on hearing aids and set to default software settings for 4 weeks.
  Interventions: Device: Hearing aid feature: Frequency Compression
- FC activated and set to hearing loss (Experimental): Frequency Compression feature activated on hearing aids and set to hearing loss cut-off for 4 weeks
  Interventions: Device: Hearing aid feature: Frequency Compression

INTERVENTIONS:
Device: Hearing aid feature: Frequency Compression — FC Deactivated/Activated & set to default/Activated & set to hearing loss
  Other Names: Non-linear Frequency Compression

SUMMARY:
The purpose of this study is to investigate the functional benefits of frequency compression vs no frequency compression or fitted to hearing loss in severe-profound hearing impaired adults with high frequency hearing losses. Thus, assessing whether hearing aids for this patient population can be adapted to improve speech perception.

DETAILED DESCRIPTION:
Frequency compression is a feature available on some digital hearing aids, which is aimed at increasing the audibility of high frequency sounds. It works by taking sounds above a fixed start frequency and compresses it into lower frequencies where residual hearing is better.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be over 18 years of age- This study is looking at the use of frequency compression & its effects of speech perception in adults.
2. No ear surgery that would make it impossible to fit a hearing aid- To ensure limited confounding variables.
3. No history of ear surgery within the last 12 months- To ensure limited confounding variables.
4. No history of ear infection(s) within the last 6 months- To ensure no contraindications and limited confounding variables to testing.
5. No otoscopic abnormality making it impossible to fit a hearing aid- To ensure no contraindications to testing.
6. Bilateral severe-profound hearing impairment with air conduction thresholds >71dBHL within the frequency range of 250Hz to 4 kHz- To analyse the effects of frequency compression on speech perception within this patient population.
7. Post lingual deafness, with good spoken English- To ensure reliability of speech testing.
8. Previous bilateral digital hearing aid experience (6+ months)- To ensure limited confounding variables.
9. Written consent required.

Exclusion Criteria:

1. Participants under the age of 18 years.
2. History of ear surgery making it impossible to fit a hearing aid.
3. History of ear surgery within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
CHEAR Auditory Perception Test | 4 weeks post hearing aid fitting with adapted hearing aid feature
  Aided Monosyllabic Speech Test
Adaptive Bamford-Kowal-Bench Test | 4 weeks post hearing aid fitting with adapted hearing aid feature
  Aided Sentence Test

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Vickers, Phd, Study Chair — UCL Ear Institute

IPD SHARING:
Plan to Share IPD: Undecided